CLINICAL TRIAL: NCT04025879
Title: A Phase 3, Randomized, Double-blind Study of Neoadjuvant Chemotherapy Plus Nivolumab Versus Neoadjuvant Chemotherapy Plus Placebo, Followed by Surgical Resection and Adjuvant Treatment With Nivolumab or Placebo for Participants With Resectable Stage II-IIIB Non-small Cell Lung Cancer
Brief Title: A Study of Neoadjuvant Chemotherapy Plus Nivolumab Versus Neoadjuvant Chemotherapy Plus Placebo, Followed by Surgical Removal and Adjuvant Treatment With Nivolumab or Placebo for Participants With Surgically Removable Early Stage Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CA209-77T; 2019-000262-38 (EudraCT Number)
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-01

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Carboplatin; Cisplatin; Paclitaxel; Pemetrexed; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neoadj. Nivo+ Pt-based Doublet Chemo followed by Adj. Nivo (Experimental)
  Interventions: Biological: Nivolumab; Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Docetaxel
- Neoadj. Plac. + Pt-based Doublet Chemo followed by Adj.Plac. (Placebo Comparator)
  Interventions: Drug: Carboplatin; Drug: Cisplatin; Drug: Paclitaxel; Drug: Pemetrexed; Drug: Placebo; Drug: Docetaxel

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: Opdivo, BMS936558
  Arms: Neoadj. Nivo+ Pt-based Doublet Chemo followed by Adj. Nivo
Drug: Carboplatin — Specified dose on specified days
Drug: Cisplatin — Specified dose on specified days
Drug: Paclitaxel — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Placebo — Specified dose on specified days
  Arms: Neoadj. Plac. + Pt-based Doublet Chemo followed by Adj.Plac.
Drug: Docetaxel — Specified dose on specified days

SUMMARY:
The main purpose of the study is to examine if periadjuvant (neoadjuvant, then adjuvant) immunotherapy will prolong event free survival in participants with early stage non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with suspected or histologically confirmed Stage IIA (> 4 cm) to IIIB (T3N2) non-small cell lung carcinoma (NSCLC) with disease that is considered resectable
* No brain metastasis
* Treatment-naive for NSCLC (no prior systemic anti-cancer treatment)
* Ability to provide surgical or biopsy tumor tissue for biomarkers
* Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1

Exclusion Criteria:

* Participants with an active, known or suspected autoimmune disease
* Any positive test for hepatitis B virus or hepatitis C virus or human immunodeficiency virus (HIV)
* Any previous anti-cancer treatment including cytotoxic, IO treatment, targeted agents, or radiotherapy for NSCLC
* Prior treatment with any anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways

Other protocol-defined inclusion/exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2023-07-26 (Actual); Study Completion 2027-07-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (106):
- United States (15):
  - Local Institution - 0104, Tampa, Florida
  - Local Institution - 0040, Atlanta, Georgia
  - Local Institution - 0120, Augusta, Georgia
  - Local Institution - 0145, Chicago, Illinois
  - Local Institution - 0078, Chicago, Illinois
  - Local Institution - 0121, Orland Park, Illinois
  - Rcca Md Llc, Bethesda, Maryland
  - Local Institution - 0076, Boston, Massachusetts
  - Local Institution - 0074, Newton, Massachusetts
  - Local Institution - 0086, Traverse City, Michigan
  - Local Institution - 0100, Lebanon, New Hampshire
  - Local Institution - 0055, Cincinnati, Ohio
  - Local Institution - 0102, Cleveland, Ohio
  - Local Institution - 0054, Houston, Texas
  - Local Institution - 0103, Fredericksburg, Virginia
- Argentina (4):
  - Local Institution - 0032, Ciudad Autonoma Beunos Aires, Buenos Aires
  - Local Institution - 0031, ABB, Buenos Aires F.D.
  - Local Institution - 0043, Buenos Aires
  - Local Institution - 0030, CABA
- Australia (4):
  - Local Institution - 0020, Sydney, New South Wales
  - Local Institution - 0033, Heidelberg, Victoria
  - Local Institution - 0122, Melbourne, Victoria
  - Local Institution - 0023, North Ballarat, Victoria
- Belgium (3):
  - Local Institution - 0002, Edegem
  - Local Institution - 0005, Liège
  - Local Institution - 0001, Roeselare
- Brazil (5):
  - Local Institution - 0035, Belo Horizonte, Minas Gerais
  - Local Institution - 0029, Ijuí, Rio Grande do Sul
  - Local Institution - 0036, São Paulo, São Paulo
  - Local Institution - 0034, São Paulo, São Paulo
  - Local Institution - 0106, São Paulo
- Local Institution - 0062, Oshawa, Ontario, Canada
- China (14):
  - Local Institution - 0115, Beijing, Beijing Municipality
  - Local Institution - 0096, Beijing, BEI
  - Local Institution - 0137, Fuzhou, Fujian
  - Local Institution - 0136, Fuzhou, Fujian
  - Local Institution - 0151, Hubei Sheng, Hubei
  - Local Institution - 0092, Changsha, Hunan
  - Local Institution - 0093, Changsha, Hunan
  - Local Institution - 0091, Changsha, Hunan
  - Local Institution - 0098, Shanghai, Shanghai Municipality
  - Local Institution - 0165, Shanghai, Shanghai Municipality
  - Local Institution - 0113, Shanghai, Shanghai Municipality
  - Local Institution - 0088, Chengdu, Sichuan
  - Local Institution - 0099, Hangzhou, Zhejiang
  - Local Institution - 0095, Shanghai
- Czechia (2):
  - Local Institution - 0041, Prague
  - Local Institution - 0042, Prague
- France (7):
  - Local Institution - 0073, Besançon
  - Local Institution - 0037, La Tronche
  - Local Institution - 0050, Montpellier
  - Local Institution - 0038, Paris
  - Local Institution - 0051, Paris
  - Local Institution - 0083, Rennes
  - Local Institution - 0146, Rouen
- Germany (12):
  - Local Institution - 0109, Immenstadt im Allgäu, Bavaria
  - Local Institution - 0110, Cologne, North Rhine-Westphalia
  - Local Institution - 0085, Berlin
  - Local Institution - 0065, Frankfurt
  - Local Institution - 0072, Georgsmarienhütte
  - Local Institution - 0071, Hamm
  - Local Institution - 0108, Heidelberg
  - Local Institution - 0064, Löwenstein
  - Local Institution - 0147, Ludwigsburg
  - Local Institution - 0063, Lübeck
  - Local Institution - 0070, Moers
  - Local Institution - 0066, München
- Local Institution - 0016, Dublin, Ireland
- Italy (3):
  - Local Institution - 0024, Forlì
  - Local Institution - 0026, Milan
  - Local Institution - 0025, Parma
- Japan (15):
  - Local Institution - 0135, Nagoya, Aichi-ken
  - Local Institution - 0124, Kashiwa-shi, Chiba
  - Local Institution - 0129, Kitakyushu-shi, Fukuoka
  - Local Institution - 0127, Kobe, Hyōgo
  - Local Institution - 0144, Kanazawa, Ishikawa-ken
  - Local Institution - 0125, Yokohama, Kanagawa
  - Local Institution - 0131, Sendai, Miyagi
  - Local Institution - 0126, Sakai-shi, Osaka
  - Local Institution - 0130, Kitaadachigun, Saitama
  - Local Institution - 0142, Bunkyo-ku, Tokyo
  - Local Institution - 0133, Bunkyo-ku, Tokyo
  - Local Institution - 0143, Chuo-ku, Tokyo
  - Local Institution - 0134, Chuo-ku, Tokyo
  - Local Institution - 0132, Fukushima
  - Local Institution - 0128, Hiroshima
- Mexico (3):
  - Local Institution - 0077, Guadalajara, Jalisco
  - Local Institution - 0027, Monterrey, Nuevo León
  - Local Institution - 0028, Chihuahua City
- Netherlands (2):
  - Local Institution - 0004, Groningen
  - Local Institution - 0003, Rotterdam
- Local Institution - 0049, Krakow, Lesser Poland Voivodeship, Poland
- Local Institution - 0117, Hato Rey, Puerto Rico
- Romania (3):
  - Local Institution - 0013, Cluj-Napoca, Cluj
  - Local Institution - 0011, Bucharest
  - Local Institution - 0012, Floreşti
- Russia (2):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
- Spain (3):
  - Local Institution - 0046, Madrid
  - Local Institution - 0044, Majadahonda - Madrid
  - Local Institution - 0045, Valencia
- Taiwan (4):
  - Local Institution - 0149, Kaohsiung City
  - Local Institution - 0119, Kaohsiung City
  - Local Institution - 0116, New Taipei City
  - Local Institution - 0112, Taipei
- Local Institution - 0007, Taunton, United Kingdom

REFERENCES:
- [Derived] Provencio M, Awad MM, Spicer JD, Janssens A, Moiseyenko F, Gao Y, Watanabe Y, Alexandru A, Guisier F, Frost N, Franke F, Hiltermann TJN, He J, Tanaka F, Lu S, Coronado Erdmann C, Sathyanarayana P, Tran P, Devas V, Cascone T. Clinical outcomes with perioperative nivolumab by nodal status in patients with stage III resectable NSCLC: phase 3 CheckMate 77T exploratory analysis. Nat Cancer. 2026 Jan;7(1):169-181. doi: 10.1038/s43018-025-01104-z. Epub 2026 Jan 8. PMID 41507539
- [Derived] Tanaka F, Watanabe Y, Sugawara S, Okami J, Muto S, Okada M, Horio Y, Tsuboi M, Sato Y, Takamochi K, Horinouchi H, Tambo Y, Seike M, Okishio K, Coronado Erdmann C, Sathyanarayana P, Meadows-Shropshire S, Ito H. Perioperative Nivolumab in Resectable Non-Small Cell Lung Cancer: A Subanalysis of Japanese Patients From CheckMate 77T. Cancer Sci. 2025 Dec 23. doi: 10.1111/cas.70300. Online ahead of print. PMID 41431434
- [Derived] Cascone T, Awad MM, Spicer JD, He J, Lu S, Sepesi B, Tanaka F, Taube JM, Cornelissen R, Havel L, Karaseva N, Kuzdzal J, Petruzelka LB, Wu L, Pujol JL, Ito H, Ciuleanu TE, de Oliveira Muniz Koch L, Janssens A, Alexandru A, Bohnet S, Moiseyenko FV, Gao Y, Watanabe Y, Coronado Erdmann C, Sathyanarayana P, Meadows-Shropshire S, Blum SI, Provencio Pulla M; CheckMate 77T Investigators. Perioperative Nivolumab in Resectable Lung Cancer. N Engl J Med. 2024 May 16;390(19):1756-1769. doi: 10.1056/NEJMoa2311926. PMID 38749033
- [Derived] Leal TA, Ramalingam SS. Neoadjuvant therapy gains FDA approval in non-small cell lung cancer. Cell Rep Med. 2022 Jul 19;3(7):100691. doi: 10.1016/j.xcrm.2022.100691. PMID 35858590
- [Derived] Hong WX, Sagiv-Barfi I, Czerwinski DK, Sallets A, Levy R. Neoadjuvant Intratumoral Immunotherapy with TLR9 Activation and Anti-OX40 Antibody Eradicates Metastatic Cancer. Cancer Res. 2022 Apr 1;82(7):1396-1408. doi: 10.1158/0008-5472.CAN-21-1382. PMID 35135810
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab + SOC Chemotherapy: Nivolumab 360 mg Q3W + SOC platinum-based doublet chemotherapy Q3W x 4 cycles as neoadjuvant treatment followed by surgery; then post surgery nivolumab 480 mg Q4W adjuvant treatment for up to 13 cycles (approximately 1 year)
- Placebo + SOC Chemotherapy: Placebo Q3W + SOC platinum-based doublet chemotherapy Q3W x 4 cycles as neoadjuvant treatment followed by surgery, then post-surgery placebo Q4W for up to 13 cycles (approximately 1 year).
Period: Randomization
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Started | 229 | 232
Completed (Continued to treatment period) | 228 | 230
Not Completed | 1 | 2
Not completed — Participant withdrew consent | 0 | 1
Not completed — Participant no longer met study criteria | 1 | 1
Period: Treatment
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Started | 228 | 230
Neoadjuvant Treatment | 228 | 230
Adjuvant Treatment | 142 | 152
Completed | 85 | 92
Not Completed | 143 | 138
Not completed — Ongoing treatment | 10 | 8
Not completed — Disease progression/recurrence | 36 | 72
Not completed — Study drug toxicity | 36 | 13
Not completed — Death | 2 | 0
Not completed — Adverse event unrelated to study drug | 21 | 14
Not completed — Participant request to discontinue study treatment | 16 | 8
Not completed — Participant withdrew consent | 1 | 3
Not completed — Participant no longer meets study criteria | 3 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other reasons | 15 | 17
Not completed — Administrative reason by sponsor | 0 | 1
Not completed — Not reported | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy | Total
Number analyzed (Participants) | 229 | 232 | 461
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 102 | 100 | 202
  >=65 years | 127 | 132 | 259
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (7.9) | 64.6 (8.4) | 64.4 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 72 | 134
  Male | 167 | 160 | 327
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 17 | 26
  Not Hispanic or Latino | 128 | 113 | 241
  Unknown or Not Reported | 92 | 102 | 194
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 66 | 50 | 116
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 155 | 175 | 330
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Event-Free Survival (EFS) by BICR
Description: The length of time from randomization to any of the following events: progression of disease or worsening of disease precluding surgery, if surgery is attempted but gross resection is abandoned due to unresectable tumor or worsening of disease, progression or recurrence of disease after surgery, progression or recurrence of disease without surgery, or death due to any cause. Progression/recurrence will be assessed by BICR per RECIST 1.1. Participants who do not undergo surgery for reason other than progression will be considered to have an event at RECIST 1.1 progression or death
Time Frame: From randomization to disease progression, worsening, recurrence, or death due to any cause (up to approximately 44 months)
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 229 | 232
Months | NA [28.94 to NA] — Insufficient number of participants with events | 18.43 [13.63 to 28.06]
Statistical Analysis 1: Comparison: Nivolumab + SOC Chemotherapy vs Placebo + SOC Chemotherapy; Test type: Superiority; p = 0.00025, Log Rank; Cox Proportional Hazard = 0.58, 95% CI 2-sided [0.43 to 0.78] — Stratified by randomization stratification factors: PD-L1 Status (>=1% vs <1%/not evaluable/indeterminate), disease stage (II vs III), histology (squamous vs non-squamous)

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time between the date of randomization and the date of death due to any cause. OS will be censored on the last date a subject was known to be alive.
Time Frame: From randomization and the date of death due to any cause.
Reporting Status: Not Posted, anticipated posting 2025-09

3. Secondary Outcome: Pathologic Complete Response (pCR) Rate
Description: Pathologic complete response (pCR) rate is defined as the percentage of randomized participants with absence of residual viable tumor in lung and lymph nodes as evaluated by blinded independent pathology review (BIPR).
Time Frame: From randomization up to approximately 44 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 229 | 232
Percentage of Participants | 25.3 [19.8 to 31.5] | 4.7 [2.4 to 8.3]
Statistical Analysis 1: Comparison: Nivolumab + SOC Chemotherapy vs Placebo + SOC Chemotherapy; Test type: Superiority; DIFFERENCE OF PCR = 20.5, 95% CI 2-sided [14.3 to 26.6] — Strata adjusted difference based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 2: Comparison: Nivolumab + SOC Chemotherapy vs Placebo + SOC Chemotherapy; Test type: Superiority; Odds Ratio (OR) = 6.64, 95% CI 2-sided [3.40 to 12.97] — Strata adjusted odds ratio using Mantel-Haenszel method

4. Secondary Outcome: Major Pathological Response (MPR) Rate
Description: Major pathological response (MPR) rate is defined as the percentage of randomized participants with ≤10% residual viable tumor in lung and lymph nodes as evaluated by blinded independent pathology review (BIPR).
Time Frame: From randomization up to approximately 44 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 229 | 232
Percentage of participants | 35.4 [29.2 to 41.9] | 12.1 [8.2 to 17.0]
Statistical Analysis 1: Comparison: Nivolumab + SOC Chemotherapy vs Placebo + SOC Chemotherapy; Test type: Superiority; DIFFERENCE OF MPR = 23.2, 95% CI 2-sided [15.8 to 30.6] — Strata adjusted difference based on Cochran-Mantel-Haenszel (CMH) method of weighting
Statistical Analysis 2: Comparison: Nivolumab + SOC Chemotherapy vs Placebo + SOC Chemotherapy; Test type: Superiority; Odds Ratio (OR) = 4.01, 95% CI [2.48 to 6.49] — Strata adjusted odds ratio using Mantel-Haenszel method

5. Secondary Outcome: The Number of Participants With Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
Time Frame: From first treatment to 30 days after last treatment of study therapy including definitive surgery and radiotherapy (up to approximately 28 months)
Population: All participants who received at least one dose of study medication in neoadjuvant or adjuvant setting.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 228 | 230
Participants | 222 | 225

6. Secondary Outcome: The Number of Participants With Serious Adverse Events (SAEs)
Description: Serious Adverse Event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is an important medical event.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of study medication in neoadjuvant or adjuvant setting.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 228 | 230
Participants | 96 | 71

7. Secondary Outcome: The Number of Participants With Select Adverse Events (AEs)
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment.
  Select AEs include endocrinopathies, diarrhea/colitis, hepatitis, pneumonitis, interstitial nephritis, and rash. Multiple event terms that may describe each of these were grouped into endocrine, GI, hepatic, pulmonary, renal, and skin select AE categories, respectively. Hypersensitivity/infusion reactions were analyzed along with the select AE categories.
Time Frame: as for outcome 5
Population: All participants who received at least one dose of study medication in neoadjuvant or adjuvant setting.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
Number analyzed (Participants) | 228 | 230
Participants
  Gastrointestinal Event | 37 | 37
  Hepatic Event | 46 | 31
  Pulmonary Event | 17 | 8
  Renal Event | 34 | 18
  Skin Event | 71 | 53
  Hypersensitivity/Infusion Reaction Event | 15 | 14
  Endocrine Event | 42 | 13

ADVERSE EVENTS:
Time Frame: All-cause mortality was assessed from randomization to primary completion (up to approximately 44 months). SAEs and Other AEs were assessed from first dose to 100 days following last dose (up to approximately 30 months)
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Arm/Group | Nivolumab + SOC Chemotherapy | Placebo + SOC Chemotherapy
All-Cause Mortality (participants affected / at risk) | 40/229 | 48/232
Serious Adverse Events (participants affected / at risk) | 109/228 | 83/230
Other Adverse Events (participants affected / at risk) | 214/228 | 212/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + SOC Chemotherapy (N=228) | Placebo + SOC Chemotherapy (N=230)
Anaemia (Blood and lymphatic system disorders) | 1 | 4
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Myelosuppression (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 4
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Immune-mediated myocarditis (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenal disorder (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 0 | 1
Immune-mediated hypophysitis (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 4 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 3
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Dehiscence (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 2 | 0
Inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Sudden death (General disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 3 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 4 | 2
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 2 | 2
Encephalomyelitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Herpetic radiculopathy (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Infectious pleural effusion (Infections and infestations) | 0 | 2
Liver abscess (Infections and infestations) | 0 | 1
Myelitis (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 3 | 0
Pneumonia (Infections and infestations) | 9 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 1
Post procedural infection (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Prostate infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 1 | 0
Rectal abscess (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Septic shock (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Systemic infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 2 | 0
Wound infection (Infections and infestations) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 1
Iatrogenic injury (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 3 | 1
Platelet count decreased (Investigations) | 1 | 3
White blood cell count decreased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to abdominal wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Paget's disease of nipple (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain oedema (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Quadriplegia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Somatic symptom disorder (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 1
Nephritis (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypersensitivity pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Laryngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary air leakage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pulmonary fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 | 1
Embolism (Vascular disorders) | 0 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Vascular compression (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab + SOC Chemotherapy (N=228) | Placebo + SOC Chemotherapy (N=230)
Anaemia (Blood and lymphatic system disorders) | 93 | 73
Leukopenia (Blood and lymphatic system disorders) | 7 | 15
Neutropenia (Blood and lymphatic system disorders) | 23 | 22
Hyperthyroidism (Endocrine disorders) | 12 | 5
Hypothyroidism (Endocrine disorders) | 28 | 4
Abdominal pain (Gastrointestinal disorders) | 12 | 15
Abdominal pain upper (Gastrointestinal disorders) | 4 | 12
Constipation (Gastrointestinal disorders) | 72 | 65
Diarrhoea (Gastrointestinal disorders) | 37 | 36
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 12
Nausea (Gastrointestinal disorders) | 67 | 78
Vomiting (Gastrointestinal disorders) | 26 | 26
Asthenia (General disorders) | 24 | 25
Chest pain (General disorders) | 11 | 12
Fatigue (General disorders) | 67 | 58
Malaise (General disorders) | 14 | 16
Non-cardiac chest pain (General disorders) | 7 | 13
Oedema peripheral (General disorders) | 16 | 9
Pain (General disorders) | 16 | 10
Pyrexia (General disorders) | 25 | 15
COVID-19 (Infections and infestations) | 28 | 22
Pneumonia (Infections and infestations) | 15 | 11
Upper respiratory tract infection (Infections and infestations) | 5 | 14
Incision site pain (Injury, poisoning and procedural complications) | 12 | 14
Procedural pain (Injury, poisoning and procedural complications) | 12 | 6
Alanine aminotransferase increased (Investigations) | 26 | 13
Aspartate aminotransferase increased (Investigations) | 15 | 14
Blood alkaline phosphatase increased (Investigations) | 15 | 7
Blood creatinine increased (Investigations) | 29 | 14
Neutrophil count decreased (Investigations) | 34 | 20
Platelet count decreased (Investigations) | 20 | 17
Weight decreased (Investigations) | 15 | 18
White blood cell count decreased (Investigations) | 29 | 10
Decreased appetite (Metabolism and nutrition disorders) | 45 | 46
Hyperglycaemia (Metabolism and nutrition disorders) | 22 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 12 | 19
Hyponatraemia (Metabolism and nutrition disorders) | 16 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 20 | 18
Myalgia (Musculoskeletal and connective tissue disorders) | 18 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 | 14
Dizziness (Nervous system disorders) | 18 | 8
Dysgeusia (Nervous system disorders) | 9 | 14
Headache (Nervous system disorders) | 19 | 18
Neuropathy peripheral (Nervous system disorders) | 25 | 25
Peripheral sensory neuropathy (Nervous system disorders) | 30 | 23
Insomnia (Psychiatric disorders) | 16 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 48
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 39 | 36
Hiccups (Respiratory, thoracic and mediastinal disorders) | 19 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 59 | 64
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 16
Rash (Skin and subcutaneous tissue disorders) | 26 | 27
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 13 | 5
Hypertension (Vascular disorders) | 12 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT04025879/Prot_SAP_000.pdf